CLINICAL TRIAL: NCT00003210
Title: A Phase II Study of Recombinant Human Interleukin-12 (rhIL-12) for the Treatment of Relapsed Lymphoma and Hodgkin's Disease
Brief Title: Interleukin-12 in Treating Patients With Previously Treated Non-Hodgkin's Lymphoma or Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02264; NCI-2012-02264 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000066067; NCI-T97-0050; DM-97073 (Other: M D Anderson Cancer Center); T97-0050 (Other: CTEP); N01CM17003 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-08-13 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2013-01

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Interleukin-12 Subunit p35; Interleukin-12

ARMS (1):
- Treatment (interleukin-12) (Experimental): Patients receive interleukin-12 subcutaneously twice a week. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: recombinant interleukin-12; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: recombinant interleukin-12 — Given subcutaneously
  Other Names: cytotoxic lymphocyte maturation factor; IL-12; interleukin-12; natural killer cell stimulatory factor; Ro 24-7472
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of interleukin-12 in treating patients with previously treated non-Hodgkin's lymphoma or Hodgkin's disease. Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill lymphoma cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate of interleukin-12 in previously treated patients with non-Hodgkin's lymphoma or Hodgkin's disease.

II. To determine the in vivo regulatory effect of interleukin-12 on Fas lingand (FasL) expression on patients' peripheral blood lymphocytes.

OUTLINE: Patients are stratified according to disease characteristics: low grade non-Hodgkin's lymphoma (follicular small cleaved, follicular mixed, small lymphocytic, and variants) versus intermediate grade non-Hodgkin's lymphoma (follicular large, diffuse large, diffuse mixed, immunoblastic, peripheral T-cell, and mantle cell) versus Hodgkin's disease.

Patients receive interleukin-12 subcutaneously twice a week. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 36-105 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated non-Hodgkin's lymphoma (all histologies except lymphoblastic and Burkitt's lymphoma) or Hodgkin's disease
* Maximum of 4 previous treatment regimens
* Measurable disease
* No CNS involvement
* Performance status - Zubrod 0-1
* Performance status - Karnofsky 80-100%
* At least 12 weeks
* Platelet count at least 75,000/mm^3
* Absolute neutrophil count greater than 1500/mm^3
* Lymphocyte count greater than 500/mm^3
* Hemoglobin at least 8.0 g/dL
* Bilirubin less than 1.5 mg/dL
* SGOT/SGPT less than 2 times normal
* Creatinine no greater than 1.6 mg/dL
* Creatinine clearance at least 60 mL/min
* No severe cardiovascular disease including active ischemic heart disease, congestive heart failure, or major arrhythmias
* No severe pulmonary disease including dyspnea with moderate to severe exertion
* HIV negative
* No active infection
* Not pregnant or nursing
* Fertile patients must use adequate contraception
* No clinically significant autoimmune disease (e.g. rheumatoid arthritis)
* No clinically significant gastrointestinal bleeding or uncontrolled peptic ulcer
* No prior allogeneic bone marrow or stem cell transplant
* At least 3 weeks since prior biologic therapy for lymphoma
* At least 3 weeks since prior chemotherapy for lymphoma
* No concurrent steroid therapy
* At least 3 weeks since prior endocrine therapy for lymphoma
* At least 3 weeks since prior radiotherapy for lymphoma
* At least 2 weeks since prior surgery

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 1998-02; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 5 years
  Simon's two-stage model will be used.

SECONDARY OUTCOMES:
Toxicity as assessed by CTC version 2.0 | Up to 5 years after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anas Younes, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States